CLINICAL TRIAL: NCT06227234
Title: Evaluation of Foreign Body Airway Obstruction Interventions Through Simulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REB23-1548
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-01

CONDITIONS: Choking; Airway Obstruction
Keywords: Basic Life Support; Foreign body airway obstruction; Abdominal thrusts; Layperson; Airway Clearance Device; Lifevac; Dechoker
MeSH Terms: conditions — Airway Obstruction | interventions — Heimlich Maneuver

STUDY DESIGN:
Intervention Model Description: Investigators will conduct an open-label, crossover, mannequin, randomized controlled trial to compare two airway clearance devices (LifeVac© and Dechoker©) with traditional abdominal thrusts as choking interventions. Participants will complete all through interventions in one of 6 randomized orders.
Masking Description: Nil, however, Outcomes Assessor will be blinded to study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- LV - DC - AT (Experimental): Order: LifeVac then Dechoker then Abdominal Thrusts
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts
- LV - AT - DC (Experimental): Order: LifeVac then Abdominal Thrusts then Dechoker
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts
- DC - AT - LV (Experimental): Order: Dechoker then Abdominal Thrusts then LifeVac
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts
- DC - LV - AT (Experimental): Order: Dechoker then LifeVac then Abdominal Thrusts
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts
- AT - LV - DC (Experimental): Order: Abdominal Thrusts then LifeVac then Dechoker
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts
- AT - DC - LV (Experimental): Order: Abdominal Thrusts then Dechoker then LifeVac
  Interventions: Other: Dechoker; Other: LifeVac; Other: Abdominal Thrusts

INTERVENTIONS:
Other: Dechoker — Participants will be shown a short educational video for each intervention. A research assistant acting as an instructor will be present to answer any questions that the students have about each of the techniques.
  After training of all three techniques is complete, participants will be asked to respond to a choking scenario, using an assigned technique (the first one in their randomized order). Participants will use a mannequin (Choking Charlie, Laerdal Medical AS, Stavanger, Norway), with a simulated food bolus placed per manufacturer's directions, to complete each scenario. Participants will have up to four minutes to complete the intervention.
  Each participant will repeat the two more times so that they attempt each intervention.
Other: LifeVac — Participants will be shown a short educational video for each intervention. A research assistant acting as an instructor will be present to answer any questions that the students have about each of the techniques.
  After training of all three techniques is complete, participants will be asked to respond to a choking scenario, using an assigned technique (the first one in their randomized order). Participants will use a mannequin (Choking Charlie, Laerdal Medical AS, Stavanger, Norway), with a simulated food bolus placed per manufacturer's directions, to complete each scenario. Participants will have up to four minutes to complete the intervention.
  Each participant will repeat the two more times so that they attempt each intervention.
Other: Abdominal Thrusts — Participants will be shown a short educational video for each intervention. A research assistant acting as an instructor will be present to answer any questions that the students have about each of the techniques.
  After training of all three techniques is complete, participants will be asked to respond to a choking scenario, using an assigned technique (the first one in their randomized order). Participants will use a mannequin (Choking Charlie, Laerdal Medical AS, Stavanger, Norway), with a simulated food bolus placed per manufacturer's directions, to complete each scenario. Participants will have up to four minutes to complete the intervention.
  Each participant will repeat the two more times so that they attempt each intervention.

SUMMARY:
WHY IS THIS STUDY BEING DONE? Little is known about the best treatment for choking. New airway clearance devices like LifeVac© and Dechoker© are being sold to help a choking person. Researchers do not know how well they work compared to other techniques like abdominal thrusts or back blows.

The purpose of this research study is to see how well bystanders can use the choking techniques.

RESEARCH QUESTION Among laypersons, which FBAO intervention (abdominal thrusts, LifeVac©, or Dechoker©) results in the greatest proportion of FBAO relief within one-minute?

PARTICIPANTS Adults aged 18 years or greater.

INTERVENTIONS View a video of each choking intervention, and then complete a choking scenario where participants will try to relieve an airway obstruction on a simulation mannequin. The three interventions are: LifeVac, Dechoker, and Abdominal Thrusts. Participants will be invited back between 90-120 days to repeat the scenarios to assess retention.

DETAILED DESCRIPTION:
Foreign body airway obstructions (FBAO, choking) result in significant mortality and morbidity globally . If left untreated, individuals suffering from airway obstructions will progress to unresponsiveness and die. For the first time in decades, a novel choking intervention is being promoted. Airway clearance devices (such as LifeVac© or Dechoker©) are non-powered suction-based devices being marketed by manufacturers as a safer, easier alternative to traditional choking interventions. However, a systematic review, conducted by Dunne et al, demonstrated insufficient evidence to recommend their use in choking guidelines. Subsequently, a mannequin simulation trial by Patterson found LifeVac© to be superior to abdominal thrusts at FBAO relief within 4 minutes (odds ratio [OR] 47.32 [95%CI 5.74 - 389.40]), whereas Dechoker© was not (OR 1.22 [95% CI 0.60 - 2.47]). This study was only conducted in healthcare professionals, and the efficacy in laypersons is still unknown.

Study Objectives 1. To evaluate the relative efficacy of airway clearance devices compared to traditional interventions among laypersons.

Research Questions and Hypotheses

1. Among laypersons, which FBAO intervention (abdominal thrusts, LifeVac©, or Dechoker©) results in the greatest proportion of FBAO relief within one-minutes?

Hypothesis: LifeVac© will relieve more FBAOs within one-minute compared to abdominal thrusts and Dechoker© based on a prior mannequin study among healthcare professionals.

Methods Investigators will conduct an open-label, crossover, mannequin, randomized controlled trial to compare two ACDs (LifeVac© and Dechoker©) with traditional abdominal thrusts as FBAO interventions.

Randomization: Using OnCore randomization service to 1 of 6 intervention orders. Randomization will be performed by a researcher not involved with participant recruitment, and allocation will be concealed until enrollment using OnCore software as well.

Pre-simulation: Prior to any intervention, each participant will receive an orientation to the simulator (Choking Charlie, Laerdal Medical AS, Stavanger, Norway), environment, and the outcomes being assessed. A member of the research team will be available to answer any questions that they have prior to starting.

Intervention: Participants will be shown the manufacturer's (LifeVac© and Dechoker©) recommended short educational video for each intervention. A publicly available online instructional video, prepared by St John Ambulance, will be used for abdominal thrusts. Immediately after watching the first training video in their allocated sequence, participants will be asked to respond to a FBAO scenario, using the assigned technique. Participants will have up to four minutes to complete the intervention. All intervention attempts will be video recorded from a standardized position. Each participant will repeat the process (instructional video, followed by scenario) two more times so that they attempt each intervention. Participants will have a short break (of approximately two minutes) between each intervention.

Follow Up: All participants will be invited back between 90 - 120 days to complete the same scenario with the 3 interventions again to assess skills retention.

ELIGIBILITY:
Inclusion Criteria:

* All adult laypersons (Aged 18 years or older)
* Able to communicate in English (to sign informed consent)
* Non-

Exclusion Criteria:

* Physical disability limiting the performance/use of the interventions
* Individuals with healthcare training (e.g., physicians, nurses, paramedics, respiratory therapists or associated students)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Odds Ratio of Airway Obstruction Relief Within One-Minute | 1 minute
  This outcome will be calculated using a mixed-effect logistic regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Comparison will be made between different pairs of devices.

SECONDARY OUTCOMES:
Odds Ratio of Airway Obstruction Relief Within Four-Minutes | 4 minutes
  This outcome will be calculated using a mixed-effect logistic regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Comparison will be made between different pairs of devices.
Hazard Ratio of Time to Airway Obstruction Relief | Maximal time allotted is 4 minutes
  This outcome will be calculated using a mixed-effect Cox regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Comparison will be made between different pairs of devices.
Odds Ratio of Airway Obstruction Relief Within One-Minute (Retention Testing) | 1 minute
  This outcome will be calculated using a mixed-effect logistic regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Retention testing will occur between 90-120 days. Comparison will be made between different pairs of devices.
Odds Ratio of Airway Obstruction Relief Within Four-Minutes (Retention Testing) | 4 minutes
  This outcome will be calculated using a mixed-effect logistic regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Retention testing will occur between 90-120 days. Comparison will be made between different pairs of devices.
Hazard Ratio of Time to Airway Obstruction Relief (Retention Testing) | Maximal time allotted is 4 minutes
  This outcome will be calculated using a mixed-effect Cox regression model, after assessment for group, carryover and period effect. Time will be calculated from when the participant first touches the mannequin to the time that the simulated food bolus is expelled from the mannequin's mouth. Participants will return for re-testing of skills between 90-120 days. Comparison will be made between different pairs of devices.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request.

REFERENCES:
- [Derived] Dunne CL, Mannani N, Cirone J, Cheng A, Blanchard IE, Holroyd-Leduc J, Wilson TA, Sauro K, McRae AD. Comparison of foreign body airway obstruction interventions among laypersons: A simulation-based, crossover, randomized controlled trial. Resusc Plus. 2025 Nov 10;26:101156. doi: 10.1016/j.resplu.2025.101156. eCollection 2025 Nov. PMID 41362661